CLINICAL TRIAL: NCT02154256
Title: Increasing, Decreasing, and Stable Incentives in a Health App Aggregator Website
Brief Title: Incentive Disbursement Pattern
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: AM14I001
Record Dates: First submitted 2014-05-27; First posted 2014-06-03 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Exercise
Keywords: walking; incentives; exercise; habits
MeSH Terms: conditions — Motor Activity; Habits

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Increasing incentives (Experimental): The investigators will offer incentives to users that begin low, and get higher over time.
  Interventions: Behavioral: Increasing incentives
- Decreasing incentives (Experimental): The investigators will offer incentives to users that start high, and decrease over time.
  Interventions: Behavioral: Decreasing incentives
- Stable incentives (Experimental): The investigators will offer incentives that stay stable over time.
  Interventions: Behavioral: stable incentives
- Usual care control (No Intervention): The investigators will offer incentives that are identical to the incentives normally offered by the investigators' partner company.

INTERVENTIONS:
Behavioral: Increasing incentives — Offer incentives that increase over time.
  Arms: Increasing incentives
Behavioral: Decreasing incentives — offer incentives that decrease over time
  Arms: Decreasing incentives
Behavioral: stable incentives — offer incentives that are stable over time, but higher than usual care
  Arms: Stable incentives

SUMMARY:
This study will be a three-arm randomized, controlled trial that the investigators will run in 2014 with approximately 4,000 users of an app called Achievemint. AchieveMint rewards users with points (which can be redeemed for prizes) for every step they take. The investigators will be testing three different point-based programs designed to encourage users to build exercise habits over the course of a month: stable incentives, increasing incentives, and decreasing incentives. After the investigators' month-long intervention period, the investigators will observe users' step counts during a month-long follow-up period to test which of the investigators' habit-building programs leaves users with the best exercise habits (or the highest step counts) after they conclude.

The time frame of observation will be 8 months.

DETAILED DESCRIPTION:
Past research has shown that paying people to exercise repeatedly can create exercise habits that last long after cash incentives are removed (Charness and Gneezy, 2009; Acland and Levy, 2013). the investigators' research will examine what kind of incentive programs build long-lasting habits most effectively. Specifically, the investigators will compare the long-term effects (based on step counts in the one month after the conclusion of the investigators' intervention) of three different interventions: (1) incentives for taking steps that remain stable over the course of a month (stable incentives); (2) incentives (of equal net value) for taking steps that start low and grow larger over the course of the month (increasing incentives); and (3) incentives (of equal net value) for taking steps that start high and decrease over the course of the month (decreasing incentives). For example, during the month-long intervention, users in group (1) will receive 6x their usual points every day for each step they take; users in group (2) will receive 2x the usual points for several days, then 3x the usual points, and so on up to 10x the usual number of points; finally, group (3) will have the same incentive schedule as group (2) but in reverse - starting with a 10x multiplier and declining. The question is this: Is it better to ease people into exercise when trying to help them form a lasting habit, to start them off intensively and then ease up the pressure, or to maintain steady, constant incentives to exercise? By examining the steps taken by members of the investigators' three experimental groups in the month following the investigators' intervention, the investigators will be able to assess whether increasing, decreasing, or stable incentives are ideal for creating lasting habits after incentives are removed. The anticipated output of this project is a published research paper.

The time frame of observation will be 8 months.

ELIGIBILITY:
Inclusion Criteria:

* all users of the Achievemint app will be eligible for inclusion

Exclusion Criteria:

* all users of the Achievemint app who are in the top 30 percentiles of activity levels will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3519 (Actual)
Dates: Start 2014-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Steps walked | 8 months
  Subjects will track steps walked with pedometers. The investigators will track how many steps they take for 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L Milkman, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Bachireddy C, Joung A, John LK, Gino F, Tuckfield B, Foschini L, Milkman KL. Effect of Different Financial Incentive Structures on Promoting Physical Activity Among Adults: A Randomized Clinical Trial. JAMA Netw Open. 2019 Aug 2;2(8):e199863. doi: 10.1001/jamanetworkopen.2019.9863. PMID 31441936